CLINICAL TRIAL: NCT05756491
Title: Outpatient Hospitalization of Unaccompanied Patients at Home for Endovascular Treatment of Peripheral Arterial Disease: a Cluster Randomized Trial.
Brief Title: Outpatient Hospitalization of Unaccompanied Patients at Home for Endovascular Treatment of Peripheral Arterial Disease.
Acronym: ABALONE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2022-A01201-42
Record Dates: First submitted 2023-01-20; First posted 2023-03-06 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Peripheral Arterial Disease
Keywords: ambulatory; accompanied patient; unaccompanied patient
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Intervention Model Description: standard care: accompanied patients Remote surveillance: unaccompanied patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental: Group1 (Experimental): In group 1: 5 centers will be randomized for the inclusion of unaccompanied patients for 24 months
  Interventions: Other: 24 months of inclusion of unaccompanied patients
- Experimental: Group2 (Experimental): In group 2: 5 other centers will be randomized for the inclusion of unaccompanied patients for 18 months
  Interventions: Other: 18 months of inclusion of unaccompanied patients
- Experimental: Group3 (Experimental): In group 3: 5 other centers will be randomized for the inclusion of unaccompanied patients for 12 months
  Interventions: Other: 12 months of inclusion of unaccompanied patients
- Experimental: Group4 (Experimental): In group 4: 5 other centers will be randomized for the inclusion of unaccompanied patients for 6 months
  Interventions: Other: 6 months of inclusion of unaccompanied patients

INTERVENTIONS:
Other: 24 months of inclusion of unaccompanied patients — inclusion for 6 months of accompanied patients in conventional outpatient care (observational period) and then inclusion for 24 months of unaccompanied with remonte surveillance patients and accompanied patients (interventional period)
  Arms: Experimental: Group1
Other: 18 months of inclusion of unaccompanied patients — inclusion for 12 months of accompanied patients in conventional outpatient care (observational period) and then inclusion for 18 months of unaccompanied with remonte surveillance patients and accompanied patients (interventional period)
  Arms: Experimental: Group2
Other: 12 months of inclusion of unaccompanied patients — inclusion for 18 months of accompanied patients in conventional outpatient care (observational period) and then inclusion for 12 months of unaccompanied with remonte surveillance patients and accompanied patients (interventional period)
  Arms: Experimental: Group3
Other: 6 months of inclusion of unaccompanied patients — inclusion for 24 months of accompanied patients in conventional outpatient care (observational period) and then inclusion for 6 months of unaccompanied with remonte surveillance patients and accompanied patients (interventional period)
  Arms: Experimental: Group4

SUMMARY:
In Westernized countries, the prevalence of peripheral arterial disease (PAD) is estimated at 15-20% of subjects over 70 years of age and is increasing considerably because of the aging of the population and the increasing prevalence of diabetes and renal insufficiency. In response to this increase in incidence, vascular surgeons must develop innovative treatments that minimize the use of resources in a context of budgetary constraints, in patients who are increasingly well informed, while maintaining the safety and effectiveness of the procedures performed.

The endovascular technique has several advantages. First, it is a minimally invasive treatment, most often performed under local anesthesia. Secondly, the duration of the procedure and the length of hospitalization are reduced. In addition, the peri-operative morbidity and mortality is extremely low.

In France, for many years, public health policies have encouraged the development of outpatient hospitalization. Endovascular treatment allows the development of outpatient care. The French Society of Vascular and Endovascular Surgery (SCVE) was the first European society to publish recommendations concerning the outpatient management of endovascular treatment of PAD. These recommendations aim to promote the development of outpatient treatment by providing a framework for practitioners wishing to offer this type of management.

Concerning the patient and according to the SCVE recommendations, all types of occlusive arterial lesions of the lower limbs can be managed on an outpatient basis and only patients with severe comorbidities are excluded from this type of hospitalization. In addition, various studies have shown the safety of outpatient hospitalization for PAD. The absence of an accompanying person on the night following the procedure is considered an exclusion criterion for outpatient care.

The objective of this Stepped-wedge Cluster Randomized Controlled Trial is to increase the use of outpatient hospitalization for endovascular treatment of PAD by proposing a care pathway adapted to people without an accompanying person on the night of the procedure at home.

ELIGIBILITY:
Inclusion Criteria:

* For all patients, the inclusion criteria are:
* Patient with symptomatic PAD (Rutherford 1-5) requiring endovascular revascularization that can be performed on an outpatient basis
* Procedure listed in the Common Classification of Medical Procedures
* Patient with a good understanding of the constraints of the study
* Patient with an ASA score of 1 to 3 (stable)
* Patient registered with the social security system
* Patient living less than 1 hour by car from the care facility or from a care facility able to care for this type of patient
* Patient willing to remain hospitalized if necessary

For accompanied patients only:

- Patient does not object to the processing of his or her data

Only for isolated patients:

* Patient with free, informed and written consent
* Patient agreeing to wear the remote monitoring device at discharge from the outpatient revascularization hospitalization
* Patient agreeing to the processing of his or her personal data with the remote monitoring provider
* Patient not living in an area not served by a cell phone network (white zone)

Exclusion Criteria:

* - Disorders of hemostasis
* Acute ischemia of the lower limbs
* Patient already included in ABALONE (2nd inclusion impossible)
* Patient already included in a type 1 interventional research protocol
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2023-04-11 (Actual); Primary Completion 2026-04-11 (Estimated); Study Completion 2026-04-11 (Estimated)

PRIMARY OUTCOMES:
Outpatient Hospitalization Rate for Endovascular Treatment of PAD at the End of the Procedure Period | 30 month

SECONDARY OUTCOMES:
Number of postoperative complications requiring re-hospitalization | 1 month
Functional improvement at 1 month as assessed by the Rutherford classification | 1 month
Assessment of patient anxiety using the HAS anxiety questionnaire | pre-procedure
Assessment of patient anxiety using the HAS anxiety questionnaire | immediately after procedure
Assessment of patient anxiety using the HAS anxiety questionnaire | Day 7

CONTACTS AND LOCATIONS:
Locations (20):
- France (20):
  - Chu Jean Minjoz, Besançon
  - Centre Hospitalier de Béziers,, Béziers
  - Hopital Universitaire Ambroise Paré,, Boulogne-Billancourt
  - CHRU Cavale Blanche, Brest
  - Chu Cote de Nacre, Caen
  - Hôpital Universitaire Gabriel Montpied, Clermont-Ferrand
  - Pôle médical du Grand large,, Décines-Charpieu
  - Hopital Le Bocage,, Dijon
  - Hopital Prive Dijon Bourgogne, Dijon
  - Clinique Mutualiste Porte de L'Orient, Lorient
  - Chu de Nantes, Nantes
  - Hopital Prive Du Confluent, Nantes
  - Chu de Nice,, Nice
  - Hôpital Saint Joseph, Paris
  - Polyclinique Francheville,, Périgueux
  - Clinique de L'Europe, Rouen
  - Centre Hospitalier Yves Le Foll-, Saint-Brieuc
  - Centre Hospitalier Privé SAINT GREGOIRE, Saint-Grégoire
  - Clinique Esquirol-Saint-Hilaire,, Saint-Hilaire
  - Médipôle Lyon Villeurbanne,, Villeurbanne